CLINICAL TRIAL: NCT01304238
Title: Systematische Dokumentation Von Patienten Mit Akutem HIT-Verdacht
Brief Title: Retrospective Registry of Patients With Acute Heparin-induced Thrombocytopenia Type II
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 108745
Record Dates: First submitted 2011-01-27; First posted 2011-02-25 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Acute HIT II (Heparin-induced Thrombocytopenia Type II)
Keywords: Retrospective evaluation of patients with acute Heparin-induced Thrombocytopenia type II treated with Fondaparinux
MeSH Terms: interventions — lepirudin; danaparoid; argatroban; Fondaparinux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- lepirudin: lepirudin treated subjects
  Interventions: Drug: lepirudin
- danaparoid: danaparoid treated subjects
  Interventions: Drug: danaparoid
- argatroban: argatroban treated subjects
  Interventions: Drug: argatroban
- fondaparinux: fondaparinux treated subjects
  Interventions: Drug: fondaparinux

INTERVENTIONS:
Drug: lepirudin — lepirudin
  Groups: lepirudin
Drug: danaparoid — danaparoid
  Groups: danaparoid
Drug: argatroban — argatroban
  Groups: argatroban
Drug: fondaparinux — fondaparinux
  Groups: fondaparinux

SUMMARY:
The purpose of this retrospective registry is to collect data about patients with acute HIT II (Heparin-induced Thrombocytopenia type II) which were treated with Lepirudin, Danaparoid, Argatroban or Fondaparinux. It is a main objective of this registry to mirror the daily routine in this indication in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Acute HIT II (Heparin-induced Thrombocytopenia type II), 4T-Score
* Treatment of HIT with Lepirudin, Danaparoid, Argatroban or Fondaparinux

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with HIT
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Schindewolf M, Steindl J, Beyer-Westendorf J, Schellong S, Dohmen PM, Brachmann J, Madlener K, Potzsch B, Klamroth R, Hankowitz J, Banik N, Eberle S, Muller MM, Kropff S, Lindhoff-Last E. Use of Fondaparinux Off-Label or Approved Anticoagulants for Management of Heparin-Induced Thrombocytopenia. J Am Coll Cardiol. 2017 Nov 28;70(21):2636-2648. doi: 10.1016/j.jacc.2017.09.1099. PMID 29169470

RESULTS

PARTICIPANT FLOW:
Groups:
- Argatroban: Participants treated with argatroban after Heparin-induced thrombocytopenia Type-II (HIT II)
- Lepirudin: Participants treated with lepirudin after HIT II
- Danaparoid: Participants treated with danaparoid after HIT II
- Fondaparinux: Participants treated with fondaparinux after HIT II
- Argatroban/Fondaparinux: Participants treated with argatroban and fondaparinux after HIT II
- Danaparoid/Argatroban: Participants treated with danaparoid and argatroban after HIT II
- Danaparoid/Fondaparinux: Participants treated with danaparoid and fondaparinux after HIT II
- Danaparoid/Lepirudin: Participants treated with danaparoid and lepirudin after HIT II
- Danaparoid/Fondaparinux/Lepirudin: Participants treated with danaparoid, fondaparinux, and lepirudin after HIT II
- Argatroban/Danaparoid/Fondaparinux: Participants treated with argatroban, danaparoid, and fondaparinux after HIT II
Period: Overall Study
Arm/Group | Argatroban | Lepirudin | Danaparoid | Fondaparinux | Argatroban/Fondaparinux | Danaparoid/Argatroban | Danaparoid/Fondaparinux | Danaparoid/Lepirudin | Danaparoid/Fondaparinux/Lepirudin | Argatroban/Danaparoid/Fondaparinux
Started | 32 | 4 | 46 | 78 | 11 | 11 | 5 | 4 | 1 | 3
Completed | 32 | 4 | 46 | 78 | 11 | 11 | 5 | 4 | 1 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Argatroban | Lepirudin | Danaparoid | Fondaparinux | Argatroban/Fondaparinux | Danaparoid/Argatroban | Danaparoid/Fondaparinux | Danaparoid/Lepirudin | Danaparoid/Fondaparinux/Lepirudin | Argatroban/Danaparoid/Fondaparinux | Total
Number analyzed (Participants) | 32 | 4 | 46 | 78 | 11 | 11 | 5 | 4 | 1 | 3 | 195
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.4 (12.3) | 61.8 (13.7) | 67.8 (13.0) | 71.7 (11.4) | 71.5 (12.1) | 60.0 (14.0) | 71.0 (8.6) | 55.3 (16.0) | 56.0 (0.0) | 63.7 (7.5) | 68.5 (12.5)
Sex/Gender, Customized [Number; unit: Participants] — Gender information is missing in one participant in the lepirudin arm.
  Participants
    Female | 10 | 1 | 21 | 35 | 5 | 5 | 2 | 2 | 1 | 2 | 84
    Male | 22 | 2 | 25 | 43 | 6 | 6 | 3 | 2 | 0 | 1 | 110
Number of participants receiving the indicated heparin treatment prior to HIT II [Number; unit: participants]
  Only unfractionated heparin (UFH) | 19 | 1 | 24 | 53 | 3 | 7 | 1 | 0 | 0 | 1 | 109
  Only low molecular weight heparin (LMWH) | 2 | 1 | 10 | 3 | 1 | 0 | 3 | 2 | 1 | 1 | 24
  UFH and LMWH | 11 | 2 | 12 | 22 | 7 | 4 | 1 | 2 | 0 | 1 | 62
Number of participants receiving the indicated AT before HIT II with regard to rationale [Number; unit: participants] — Multiple responses are possible. AT, anticoagulant treatment. "Rationale" refers to the initial reason for giving antithrombotics, e.g., for prophylaxis or for therapy of thrombosis.
  participants
    Prophylactic | 24 | 2 | 39 | 66 | 9 | 8 | 2 | 3 | 0 | 2 | 155
    Therapeutic | 14 | 2 | 18 | 21 | 6 | 6 | 3 | 2 | 1 | 3 | 76
Number of participants receving the indicated AT before HIT II (specified) with regard to rationale [Number; unit: participants] — Multiple responses are possible. AT, anticoagulant treatment.
  participants
    Prophylaxis (no further specification) | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 5
    Prophylaxis: Surgery | 12 | 2 | 11 | 62 | 6 | 5 | 1 | 3 | 0 | 0 | 102
    Prophylaxis: Internal Medicine | 13 | 0 | 27 | 4 | 2 | 5 | 1 | 1 | 0 | 2 | 55
    Prophylaxis: Neurology/Neurosurgery | 2 | 0 | 10 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 14
    Indication for thromboembolic therapy | 14 | 2 | 18 | 21 | 6 | 6 | 3 | 2 | 1 | 3 | 76
Number of participants with the indicated thromboembolic therapy (specified) [Number; unit: participants] — Multiple responses are possible.
  participants
    Deep vein thrombosis | 5 | 0 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 14
    Pulmonary embolism | 4 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 0 | 1 | 12
    Peripheral artery occlusive disease | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
    Acute coronary syndrome | 1 | 1 | 3 | 4 | 0 | 2 | 0 | 1 | 0 | 0 | 12
    Alternative anticoagulation in atrial fibrillation | 4 | 0 | 9 | 13 | 1 | 0 | 2 | 0 | 0 | 2 | 31
    Alternative anticoagulation in cardiac valve | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 4
    Other | 3 | 1 | 3 | 0 | 2 | 4 | 0 | 0 | 1 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Diagnosed With Thrombosis and/or Pulmonary Embolism After the Occurrence of HIT II
Description: Thrombosis is a clotting in a blood vessel. Pulmonary embolism is a clot, usually from the deep veins of the legs, carried away with the venous bloodstream into the lungs, where it may block pulmonary vessels. Participants' medical records were used to abstract data that were collected on standardized hard copy Case Report Forms (CRFs).
Time Frame: 19 January 2005 to 25 October 2009
Population: All documented participants diagnosed with suspected acute HIT II and a 4T Score of ≥4 who had received at least one dose of argatroban, lepirudin, danaparoid, or fondaparinux. The 4T score (range: 0-8) was developed to predict the probability of HIT.
Measure: Number; unit: participants
Arm/Group | Argatroban | Lepirudin | Danaparoid | Fondaparinux | Argatroban/Fondaparinux | Danaparoid/Argatroban | Danaparoid/Fondaparinux | Danaparoid/Lepirudin | Danaparoid/Fondaparinux/Lepirudin | Argatroban/Danaparoid/Fondaparinux
Number analyzed (Participants) | 32 | 4 | 46 | 78 | 11 | 11 | 5 | 4 | 1 | 3
participants
  Thrombosis | 31 | 4 | 45 | 78 | 11 | 6 | 5 | 1 | 1 | 3
  No thrombosis or pulmonary embolism | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 2 | 0 | 0
  Pulmonary embolism | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Thrombosis and pulmonary embolism | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants Diagnosed With Bleeding After the Occurrence of HIT II
Description: Participants' medical records were used to abstract data that were collected on standardized hard copy Case Report Forms (CRFs). Bleeding was documented in the participant files.
Time Frame: 19 January 2005 to 25 October 2009
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Argatroban | Lepirudin | Danaparoid | Fondaparinux | Argatroban/Fondaparinux | Danaparoid/Argatroban | Danaparoid/Fondaparinux | Danaparoid/Lepirudin | Danaparoid/Fondaparinux/Lepirudin | Argatroban/Danaparoid/Fondaparinux
Number analyzed (Participants) | 32 | 4 | 46 | 78 | 11 | 11 | 5 | 4 | 1 | 3
participants
  No Bleeding | 30 | 4 | 43 | 74 | 11 | 8 | 5 | 2 | 1 | 3
  Bleeding | 2 | 0 | 3 | 4 | 0 | 3 | 0 | 2 | 0 | 0

3. Secondary Outcome: Number of Participants With Fatal Complications After the Occurrence of HIT II
Description: Participants' medical records were used to abstract data that were collected on standardized hard copy Case Report Forms (CRFs). A fatal complication is defined as a complication resulting in death.
Time Frame: 19 January 2005 to 25 October 2009
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Argatroban | Lepirudin | Danaparoid | Fondaparinux | Argatroban/Fondaparinux | Danaparoid/Argatroban | Danaparoid/Fondaparinux | Danaparoid/Lepirudin | Danaparoid/Fondaparinux/Lepirudin | Argatroban/Danaparoid/Fondaparinux
Number analyzed (Participants) | 32 | 4 | 46 | 78 | 11 | 11 | 5 | 4 | 1 | 3
participants
  No fatal complication | 27 | 4 | 35 | 78 | 11 | 9 | 5 | 2 | 1 | 3
  Fatal complication | 5 | 0 | 11 | 0 | 0 | 2 | 0 | 2 | 0 | 0

4. Secondary Outcome: Number of Participants Who Underwent Amputation After the Occurrence of HIT II
Description: Participants' medical records were used to abstract data that were collected on standardized hard copy Case Report Forms (CRFs).
Time Frame: 19 January 2005 to 25 October 2009
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Argatroban | Lepirudin | Danaparoid | Fondaparinux | Argatroban/Fondaparinux | Danaparoid/Argatroban | Danaparoid/Fondaparinux | Danaparoid/Lepirudin | Danaparoid/Fondaparinux/Lepirudin | Argatroban/Danaparoid/Fondaparinux
Number analyzed (Participants) | 32 | 4 | 46 | 78 | 11 | 11 | 5 | 4 | 1 | 3
participants
  No amputation | 32 | 4 | 46 | 78 | 11 | 10 | 5 | 3 | 1 | 3
  Amputation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

5. Secondary Outcome: Number of Participants Who Were Diagnosed With Thrombocytopenia (Recurrent of Persistent) After the Occurrence of HIT II
Description: Participants' medical records were used to abstract data that were collected on standardized hard copy Case Report Forms (CRFs). Thrombocytopenia after HIT-II was documented in the participant files.
Time Frame: 19 January 2005 to 25 October 2009
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Argatroban | Lepirudin | Danaparoid | Fondaparinux | Argatroban/Fondaparinux | Danaparoid/Argatroban | Danaparoid/Fondaparinux | Danaparoid/Lepirudin | Danaparoid/Fondaparinux/Lepirudin | Argatroban/Danaparoid/Fondaparinux
Number analyzed (Participants) | 32 | 4 | 46 | 78 | 11 | 11 | 5 | 4 | 3 | 1
participants
  Recurrent thrombocytopenia | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 0
  Persistent thrombocytopenia | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  No thrombocytopenia | 31 | 4 | 44 | 78 | 11 | 8 | 5 | 3 | 1 | 1

6. Secondary Outcome: Number of Participants Who Experienced Skin Changes (Erythema and Necrosis) After the Occurrence of HIT II
Description: Participants' medical records were used to abstract data that were collected on standardized hard copy Case Report Forms (CRFs). Erythema is a redness of the skin caused by hyperemia. Necrosis is the premature death of cells or tissues.
Time Frame: 19 January 2005 to 25 October 2009
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Argatroban | Lepirudin | Danaparoid | Fondaparinux | Argatroban/Fondaparinux | Danaparoid/Argatroban | Danaparoid/Fondaparinux | Danaparoid/Lepirudin | Danaparoid/Fondaparinux/Lepirudin | Argatroban/Danaparoid/Fondaparinux
Number analyzed (Participants) | 32 | 4 | 46 | 78 | 11 | 11 | 5 | 4 | 1 | 3
participants
  No skin changes | 32 | 4 | 45 | 78 | 11 | 11 | 5 | 3 | 0 | 3
  Skin changes | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical record data; thus, no assessments of serious or non-serious adverse events are possible.
Arm/Group | Argatroban | Lepirudin | Danaparoid | Fondaparinux | Argatroban/Fondaparinux | Danaparoid/Argatroban | Danaparoid/Fondaparinux | Danaparoid/Lepirudin | Danaparoid/Fondaparinux/Lepirudin | Argatroban/Danaparoid/Fondaparinux
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Due to the retrospective nature of the data collection in this study, it is impossible to be precise about dose and frequency of dosing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.